CLINICAL TRIAL: NCT06274697
Title: Validation Study of a Magnetic Sensor in Arterial Flow Recording, Compared With the Reference Method (Echodoppler), at Various Peripheral Arterial Sites
Brief Title: Validation of a Magnetic Sensor in Arterial Flow Recording, Compared With the Reference Method, at Various Peripheral Arterial Sites
Acronym: COMADO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: phymedexp (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0391; 2023-A01784-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Lower Extremity Artery Disease
Keywords: Peripheral arterial disease; Arterial Obstructive Disease; Doppler ultrasound; Magnetic sensors;
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic sensor (Experimental): The CapMagic device is a small magnetic sensor, whose technology is derived from magnetocardiography, with a very weak field identical to that of a refrigerator magnet, which is placed on the foot or toe to record curves reflecting the state of the arterial network. It does not require direct skin contact.
  Interventions: Device: Evaluation by magnetic sensor

INTERVENTIONS:
Device: Evaluation by magnetic sensor — Evaluation by magnetic sensor on arm and leg

SUMMARY:
The measurement of magnetic fields emitted by cardiac activity has already been studied in magneto-cardiography. To date, however, this technology has never been evaluated in the peripheral circulation.

The magnetic susceptibility of iron in the circulating blood and the ionic currents in the blood stream generate a very weak induced magnetic current, which can be detected by the micro-sensor of the prototype investigators wish to study.

Proving the validity of this prototype would make it a new diagnostic and even prognostic tool, non-invasive, less costly and more accessible than Doppler for screening peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the Heart-Lung Unit of the Montpellier University Hospital, for any reason whatsoever
* Patient with lower extremity artery disease (LEAD) (stage 1 to 4 according to Leriche and Fontaine) or not (absence of LEAD)
* Age ≥ 18 years

Exclusion Criteria:

* Patient with a metal implant in the vicinity of the device's area of use
* Patient requiring additional hygiene precautions
* Subject not affiliated to a social security scheme or not benefiting from such a scheme.
* Pregnant or breast-feeding woman, patient unable to give consent, protected adult, vulnerable persons
* Subject deprived of liberty by judicial or administrative decision
* Patient refusing to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of the two curve amplitudes (y) versus time (x) between the signal recording obtained by the CapMagic prototype on the radial artery and the pulsed echo-Doppler recording on the radial artery | On day 1
  Correlation of the two curve amplitudes (y) versus time (x) between the signal recording obtained by the CapMagic prototype on the radial artery and the pulsed echo-Doppler recording on the radial artery, in adult patients with or without AOMI in hospital.
  The result is expressed by a Spearman correlation coefficient ranging from -1 to 1, with 0 corresponding to no correlation and 1 corresponding to a perfect positive correlation

SECONDARY OUTCOMES:
Correlations of the two curve amplitudes (y) versus time (x) between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording, measured on the plantar artery on one side and on the pulpal artery on the other | On day 1
  Correlations of the two curve amplitudes (y) versus time (x) between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording, measured on the plantar artery on one side and on the pulpal artery on the other, in adult patients with or without LEAD in hospital.
  The result is expressed by a Spearman correlation coefficient ranging from -1 to 1, with 0 corresponding to no correlation and 1 corresponding to a perfect positive correlation
Correlation of the Pulsatility index (or Gosling Pulsatility index) between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording | On day 1
  IP=P/M where P=maximum amplitude of the trace (from highest positive value, i.e. peak systolic, to lowest value) and M=average circulatory velocity, averaged over the entire cardiac cycle. Calculated from the Doppler or CapMagic curves.
Correlation of the Systolic rise time (SRT) between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording | On day 1
  Systolic rise time (SRT), (ms) : the time between the foot and the peak of the pulse wave. Calculated from the Doppler or CapMagic curves.
Correlation of the Systolic peak between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording | On day 1
  Systolic peak, Measured in cm/s or mV: Peak height in systole. Calculated from the Doppler or CapMagic curves.
Correlation of the maximum acceleration of systolic rise between the signal recording obtained by the CapMagic prototype and the pulsed echo-Doppler recording | On day 1
  The maximum acceleration of systolic rise (cm/s2) calculated from the Doppler or CapMagic curves.
Correlation of Presence of critical ischemia measured by the CapMagic prototype and the pulsed echo-Doppler recording | On day 1
  critical ischemia is defined by systolic pressure at toe < 30 mmHg or ankle < 50mmHg, or diagnosis of critical ischemia retained by the team in the impossibility of obtaining pressure measurements

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center, Montpellier, France